CLINICAL TRIAL: NCT02401984
Title: Zürcher Adoleszenz-Screening-Instrument Psychischer Störungen
Brief Title: Zurcher Adolescent Screening for Mental Disorder
Acronym: ZASMD
Status: Completed | Type: Observational
Sponsor: Filomena Sabatella (Other)
Responsible Party: Sponsor-Investigator, Filomena Sabatella, MSc, Zurich University of Applied Sciences
Organization: Zurich University of Applied Sciences (Other)
Other Study IDs: 2014-0575
Record Dates: First submitted 2015-03-03; First posted 2015-03-30 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Mental Disorders
MeSH Terms: conditions — Mental Disorders | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Screening: A Screening tool will be administered to the participants.
  Interventions: Other: Screening

INTERVENTIONS:
Other: Screening — Participants will fill out a short screening questionnaire where different aspects of mental health and behavioral problems will be assessed.

SUMMARY:
Mental disorders are common in youth and adults. Symptoms of mental are aggravated by unemployment. Compared to the working population, the unemployed have higher rates of poor health, a tendency toward negative emotionality and depression, show symptoms of exhaustion more frequently, and experience disturbed sleep or have a sleep disorder. It can be reasonably expected that unemployment in adolescents and young adults causes the same symptoms and behaviors as in adults. In those youth with a mental disorder, particularly an untreated one, the transfer from school to the employment market can be hindered. At the same time, the investigators notice an increase in early disability pensions due to mental health issues among adolescents. Thus, the early recognition and treatment of mental disorders and psychological strain is crucial in promoting the employment of young people and supporting their connection to the employment market.With this project the investigators want to implement an early intervention and reach out to unemployed youth. The investigators identified the period between graduation and first employment as the ideal moment of intervention, because this time period is a critical period in which young people are exposed to increasing personal challenges. Conducting an intervention before a psychological stress transforms into a mental disorder, can prevent harm and suffering to the afflicted person. In addition, early intervention could help prevent the need to enroll in the early disability pension program.

DETAILED DESCRIPTION:
Mental disorders are common. A WHO study shows (Gore, Bloem, Ferguson, Coffey and Mathers, 2011) that during adolescence; most of the years lost because of illness are due to neuropsychiatric disorders such as depression, substance abuse and schizophrenia. Steinhausen, Metzke and Kannenberg (1998) found that 22% of the children and adolescents living in the canton of Zurich, suffer from mental disorders. The figures are comparable with Wittchen, Nelson and Lachner (1998) who fund 27% of the adolescents fitting the DSM IV (Diagnostic and Statistical Manual) criteria for mental disorders.

Mental disorders are particularly stressful in combination with unemployment. Unemployed are often in a worse physical condition compared to employed people; they tend to negative emotional states and depression, fatigue and sleep disorders. It is to be expected that unemployment will have the same effect on adolescents. Fergusson, Horwood and Lynskey (1997) showed that in 16 to 25 years old, the increase of the unemployment was correlated with the increase of mental distress having consequences like depression, anxiety, substance abuse and attempts to suicide.

The aim of this project is to validate a screening tool for the early recognition of mental disorders among young unemployed. The screening tool will be composed by no more than 50 items.

The participants will be requested to fill out the screening tool and in a second phase, they will be asked to participate in a face to face, standardized clinical Interview, the Munich-Composite International Diagnostic Interview (M-CIDI) (Wittchen, Lachner, Wunderlich and Pfister, 1998).

To ensure that the screening tool differentiates between 'at risk' and 'non at risk' patients, the sample will be composed by 40 unemployed young adults, Age 16-25 and 40 working young adults, age 16-25.

Statistical Analysis: After the data collection the data from the screening and the clinical interview will be tested for sensitivity and specificity. To evaluate both the Receiver Operating Characteristic (ROC) and other methods will be used. The prognostic validity of the screening tool will be additionally calculated with a logistic regression. The data analysis will be executed with SPSS 21.

Missing data will be excluded from the sample.

ELIGIBILITY:
Inclusion Criteria:

* 40 unemployed Young adults, Age 16-25,
* 40 working Young adults, Age 16-25,
* informed consent to participate in the study.

Exclusion Criteria:

* insufficient understanding of the German language.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants will be recruited in Institutions Coaching unemployed Young People.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
DSM IV diagnosis | 1-2 Week

CONTACTS AND LOCATIONS:
Overall Officials: Agnes von Wyl, Professor, Study Director — University of applied sciences
Locations (1):
- Toni Areal, Zurich, Canton of Zurich, Switzerland